CLINICAL TRIAL: NCT06830486
Title: The Effects of Cardiorespiratory Fitness, Physical Activity and Sedentary Behavior on Insulin Resistance Among Breast Cancer Survivors Being Treated With Anti-estrogen Endocrine Therapies
Brief Title: Effects of Activity on Diabetes Risk Among Breast Cancer Survivors on Endocrine Therapy (ABIDE)
Acronym: ABIDE
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3245.cc
Record Dates: First submitted 2023-12-01; First posted 2025-02-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Exercise; Breast Cancer; Endocrine Therapy; Insulin Resistance; Body Composition
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SERM: These patients are being treated with a SERM for at least one year prior to enrolling in the study.
  Interventions: Other: No intervention
- Aromatase Inhibitor: These patients are being treated with an aromatase inhibitor for at least one year prior to enrolling in the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is performed. Participants who have been treated with either a SERM or aromatase inhibitor are recruited and analyzed in separate groups, but the study design for all participants is identical.

SUMMARY:
The aim of this study is to learn more about how physical activity and cardiorespiratory fitness are related to diabetes risk among breast cancer patients prescribed an endocrine therapy.

DETAILED DESCRIPTION:
80 women between the ages of 18-80 years will be recruited for this study. The study design consists of two separate in-person visits to University of Colorado Anschutz Medical Campus or Colorado State University. The study consists of glucose testing, a body composition scan, exercise testing, and a two-week period of free living activity monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Female
* diagnosed with breast cancer
* age 18-80 years
* Completed surgery, chemo- and/or radiation therapy
* Prescribed aromatase inhibitor or SERM for at least one year from the time of screening

Exclusion Criteria:

* Age < 18 or > 80
* Type 1 diabetes
* Type 2 diabetes
* Prescribed anti-hyperglycemic medication, insulin, or sulfonylurea.
* Pregnant, breastfeeding or planning to become pregnant in next 2 months
* Have absolute contraindications to exercise testing which are:

  1. Unstable angina
  2. Recent myocardial infarction, cardiac surgery, or vascular surgery (<3 months)
  3. Uncontrolled high blood pressure
  4. Heart failure
  5. Peripheral artery disease (based on report of symptomatic claudication)
  6. Hepatic or renal disease
  7. Severe arthritis or mobility impairment that would interfere with exercise testing
* Suspected cognitive impairment that would prevent understanding or comprehension of study procedures.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female.
Study Population: Breast cancer survivors prescribed endocrine therapy for at least one year
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | Immediately after the consent form is signed
  Insulin resistance will be measured through oral glucose tolerance testing
Body Composition | Immediately after the insulin resistance measurement
  Body composition will be measured through DEXA scan
Maximal Exercise Capacity | Within 2-60 days of insulin resistance measurement
  Maximal exercise capacity measured through graded exercise test on stationary bicycle
Daily Activity | 2-60 days following insulin resistance measurement
  Daily activity measured using activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Scalzo, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University Of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided